CLINICAL TRIAL: NCT02706522
Title: Effect of Oral Carbohydrate on Serum S-100β Protein and Development of Postoperative Delirium in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, SeHee Na, Associate Professor MD, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2015-0317
Record Dates: First submitted 2016-03-02; First posted 2016-03-11 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance; Inflammation; Delirium
MeSH Terms: conditions — Insulin Resistance; Inflammation; Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allocated to Carbohydrated group (Experimental): 1. Patients was administered in hospital
  2. Randomization
  3. Patient was allocated to Carbohydrated group
  4. Patients received 400 mL of oral isotonic glucose (No NPO®, Daesang, Korea) 12 hours before anesthesia and 400 mL 2 hours before. CHL composition was standard: 12.5 g of carbohydrate per 100 mL, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 250 mOsm/kg and 50 kcal.
  Interventions: Dietary Supplement: Allocated to Carbohydrated group
- Allocated to Placebo group (Placebo Comparator): 1. Patients was administered in hospital
  2. Randomization
  3. Patient was allocated to Placebo group
  4. Patients received 400 mL of water 12 hours before anesthesia and 400 mL 2 hours before anesthesia.
  Interventions: Dietary Supplement: Allocated to Placebo group

INTERVENTIONS:
Dietary Supplement: Allocated to Carbohydrated group — Patients received 400 mL of oral isotonic glucose (No NPO®, Daesang, Korea) 12 hours before anesthesia and 400 mL 2 hours before. CHL composition was standard: 12.5 g of carbohydrate per 100 mL, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 250 mOsm/kg and 50 kcal.
  Other Names: No NPO
  Arms: Allocated to Carbohydrated group
Dietary Supplement: Allocated to Placebo group — Patients received 400 mL of oral flavored water (Placebo) 12 hours before anesthesia and 400 mL 2 hours before
  Other Names: flavored water
  Arms: Allocated to Placebo group

SUMMARY:
This study is to evaluate the effects of preoperative carbohydrate intake on perioperative neuroinflammation and development of delirium.

DETAILED DESCRIPTION:
Perioperative insulin resistance may primarily contribute to development of postoperative delirium in high risk patients. Preoperative administration of oral carbohydrate reduces insulin resistance. The investigators aimed to investigate the influence of carbohydrate loading on the serum level of S-100β, a surrogate marker of delirium, and the incidence of postoperative delirium in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip replacement or total knee replacement surgery

Exclusion Criteria:

* Diabetes
* Dementia
* Gastro-esophageal reflux
* Upper gastrointestinal motility disorder
* Inflammatory bowel disease
* Intraperitoneal malignancy history
* Inability to perform cognitive function test

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
serum S-100β level | Postoperative 1 hr

IPD SHARING:
Plan to Share IPD: No